CLINICAL TRIAL: NCT02967133
Title: Nivolumab With or Without Nab-Paclitaxel in Previously Treated, Advanced Stage, Non-small Cell Lung Cancer: A Randomized Phase II Study
Brief Title: A Study of Nivolumab +/- Nab-paclitaxel in Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Celgene Corporation (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-31
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Results first posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-08

CONDITIONS: Non-Small-Cell Lung Cancer Metastatic; Non-Small Cell Carcinoma of Lung, TNM Stage 4; Nonsmall Cell Lung Cancer; Non Small Cell Lung Cancer Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator): Nivolumab q 14 days until disease progression/toxicity
  Interventions: Drug: Nivolumab
- Arm B (Active Comparator): Nivolumab every 21 days until disease progression
  Nab-paclitaxel every 21 days
  Interventions: Drug: Nivolumab; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Nivolumab — Arm A: Nivolumab 240 mg via intravenous infusion (IV) over 30 minutes day 1 of each 14 day cycle until disease progression or not tolerated.
  Arm B: Nivolumab 360 mg via intravenous infusion (IV) over 30 minutes day 1 of every 21 day treatment cycle until progression or not tolerated.
  Other Names: Opdivo
Drug: nab-paclitaxel — Patients in arm B receive nab-paclitaxel at a dose of 100 mg/m2 over intravenous infusion on Days 1 and 8 of each 21 day cycle.
  Other Names: abraxane
  Arms: Arm B

SUMMARY:
The optimal prioritization of second-line chemotherapy and immune therapy based on demographic or biomarker data is an area of ongoing investigation. The hypothesis of this study is that there may be an additive or synergistic antitumor effect of combined chemotherapy and nivolumab in the second-line treatment of NSCLC as an important concept to test in a clinical trial. Previously treated NSCLC remains a setting of unmet clinical need despite recent clinical research progress. Early progression for a subset of NSCLC patients receiving nivolumab is a specific area of clinical need.

DETAILED DESCRIPTION:
Nab-paclitaxel will be added to standard nivolumab therapy in previously treated advanced stage non-small cell lung cancer to help prevent early progression and to improve progression free survival. The primary endpoint will be to determine if the addition of nab-paclitaxel to nivolumab improves progression free survival compared to nivolumab alone. Retrospective studies will be conducted to analyze blood based immune biomarkers, and tumor biomarkers to better understand the effect that nivolumab combined with chemotherapy has on the immune system in NSCLC. Patients with advanced stage non-small cell lung cancer who have progression of cancer after receiving platinum doublet chemotherapy will be randomized to receive nivolumab with or without nab-paclitaxel. Patients on both arms will receive a maximum of one year of therapy with the option to retreat at progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, Stage IV non-small cell lung cancer (per the Union Internationale contre le Cancer/American Join Committee on Cancer staging system, 7th edition) or recurrent incurable non-small cell lung cancer that has progressed after first-line chemotherapy.
2. Prior Therapy: Platinum doublet chemotherapy for current diagnosis of advanced lung cancer. Only one prior line of chemotherapy for advanced lung cancer allowed. Adjuvant chemotherapy, neoadjuvant chemotherapy, or chemoradiotherapy given for early stage lung cancer at least 6 months prior to diagnosis of recurrent/metastatic disease is not counted as a line of therapy for advanced lung cancer. Patients who received platinum doublet therapy with or without radiotherapy as part of treatment for early stage non-small cell lung cancer less than 6 months after developing stage 4 or recurrent incurable disease will be considered study eligible by the criterion of having received one line of chemotherapy for non-small cell lung cancer.
3. EGFR, ALK and ROS biomarker positive tumors are eligible as long as the patient has received at least one standard oral, molecular inhibitor therapy in addition to standard platinum doublet chemotherapy. More than one molecular inhibitor is allowed such as a first generation EGFR inhibitor followed by a next generation EGFR inhibitor when T790 mutation develops. Prior molecular therapy for biomarker positive tumors such as (but not limited to) MET, RET and BRAF allowed but not required.
4. Prior chemotherapy must have been completed 21 days prior to initiation of protocol therapy and all toxicities must < grade 2.
5. Patients must have < Grade 2 or pre-existing neuropathy (per CTCAE).
6. Palliative radiation must have been completed 2 weeks prior to the initiation of study therapy.
7. All patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20mm with conventional techniques or as ≥10mm with spiral CT scan.
8. ECOG Performance Status: 0-1
9. Second malignancy: No "currently active" second malignancy other than non-melanoma skin cancers.
10. Brain metastases: brain metastases must have been treated at least 2 weeks prior to enrollment, be asymptomatic from brain metastases, stable on brain imaging, and not be receiving a supra-physiologic dose of steroids (> 10 mg prednisone daily or equivalent).
11. Non-pregnant and non-nursing. The effect of nab-paclitaxel and nivolumab on the fetus is unknown.
12. Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses > 1 year.
13. Male patients must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.
14. Age ≥18 years.
15. Required Initial Laboratory Values:

    Leukocytes ≥2000/ µl Hemoglobin >9.0 g/dL Platelets ≥100,000/ µl ANC ≥1,500/mcL

    Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

    Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL

    Male CrCl = (140 - age in years) x weight in kg x 1.00

    Total Bilirubin <1.5 mg/dl (except for subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dl) SGOT (AST) <2.5 x ULN ALP <2.5 x ULN in absence of liver metastases (<5 x ULN if liver metastases present PTT <1.5 x ULN
16. An archival tumor sample from either a prior core needle biopsy or surgical specimen must be available to be submitted for correlative studies as an eligibility requirement prior to registration. The sample must be shipped within 6 weeks of enrollment. Participants without an available archival tumor sample are considered ineligible.

Exclusion Criteria:

1. Prior nab-paclitaxel chemotherapy excluded.
2. Prior immune therapy for NSCLC excluded. Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
3. Patients will be excluded if they have an active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
4. Patients will be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10mg/day prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence or active autoimmune disease.
5. Patients should be excluded if they test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
6. Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
7. Allergies and Adverse Drug Reaction: History of allergy to study drug components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bertagnolli, MD, Principal Investigator — Alliance Foundation Trials, LLC.; Neal Ready, MD, PhD, Study Chair — Alliance Foundation Trials, LLC.
Locations (4):
- United States (4):
  - St. Elizabeth's Healthcare, Edgewood, Kentucky
  - Metro Minnesota community oncology research consortium, Saint Louis Park, Minnesota
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized (de-identified) data generated from biospecimens used for future correlative research, including somatic and constitutional (germline) genomic data, may be shared with other researchers or deposited in a publicly accessible or controlled-access data repositories. Correlative study results and data will never be returned to individual patients.

REFERENCES:
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Socinski MA, Bondarenko I, Karaseva NA, Makhson AM, Vynnychenko I, Okamoto I, Hon JK, Hirsh V, Bhar P, Zhang H, Iglesias JL, Renschler MF. Weekly nab-paclitaxel in combination with carboplatin versus solvent-based paclitaxel plus carboplatin as first-line therapy in patients with advanced non-small-cell lung cancer: final results of a phase III trial. J Clin Oncol. 2012 Jun 10;30(17):2055-62. doi: 10.1200/JCO.2011.39.5848. Epub 2012 Apr 30. PMID 22547591
- [Background] Liu Z, Wei Z, Hu Y, Gao F, Hao L, Fang P, Sun S, Li J, Jiao S. A phase II open-label clinical study of comparing nab-paclitaxel with pemetrexed as second-line chemotherapy for patients with stage IIIB/IV non-small-cell lung cancer. Med Oncol. 2015 Aug;32(8):216. doi: 10.1007/s12032-015-0660-5. Epub 2015 Jul 14. PMID 26168982
- [Background] Camidge R. et al. ORAL02.05 Safety and Efficacy of First-Line Nivolumab (NIVO; Anti-Programmed Death-1 [PD-1]) and Ipilimumab in Non-Small Cell Lung Cancer (NSCLC) World Lung Cancer Meeting, Denver, CO September 2015.
- [Background] Adams S, et al. OT1-01-06 A phase III randomized trial of atezolizumab in combination with nab-paclitaxel as first line therapy for patients with metastatic triple-negative breast cancer (mTNBC) San Antonio Breast Cancer Meeting, San Antonio, TX December 2015.
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Freidlin B, Korn EL, George SL. Data monitoring committees and interim monitoring guidelines. Control Clin Trials. 1999 Oct;20(5):395-407. doi: 10.1016/s0197-2456(99)00017-3. PMID 10503800
- [Background] Kaplan, E.L., Meier, P., Nonparametric estimation from incomplete observations. J Am Stat Assoc, 1958. 53(282): p. 457-481.
- [Background] Mantel N. Evaluation of survival data and two new rank order statistics arising in its consideration. Cancer Chemother Rep. 1966 Mar;50(3):163-70. No abstract available. PMID 5910392
- [Background] Cox, D.R. Regression models and life-tables. J R Stat Soc 1972 34: p.187-220.
- [Background] Fine, J., Gray R., A proportional hazards model for the sub distribution of a competing risk. J Am Stat Assoc, 1999. 94: p. 496-509.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Nivolumab Alone): Nivolumab q 14 days until disease progression/toxicity Nivolumab: Arm A: Nivolumab 240 mg via intravenous infusion (IV) over 30 minutes day 1 of each 14 day cycle until disease progression or not tolerated.
- Arm B (Nivolumab + Nab-Paclitaxel): Nivolumab every 21 days until disease progression Nab-paclitaxel every 21 days nab-paclitaxel: Patients in arm B receive nab-paclitaxel at a dose of 100 mg/m2 over intravenous infusion on Days 1 and 8 of each 21 day cycle.
Period: Overall Study
Arm/Group | Arm A (Nivolumab Alone) | Arm B (Nivolumab + Nab-Paclitaxel)
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Nivolumab Alone) | Arm B (Nivolumab + Nab-Paclitaxel) | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 71] | 70.5 [68 to 82] | 69 [54 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: This study will compare the progression-free survival of patients with advanced stage non-small cell lung cancer whose cancer has progressed after standard first-line platinum based doublet chemotherapy is improved with nivolumab plus nab-paclitaxel compared to nivolumab alone. A progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: 13 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Nivolumab Alone) | Arm B (Nivolumab + Nab-Paclitaxel)
Number analyzed (Participants) | 3 | 4
Months | 1.3 [1.0 to NA] — Insufficient number of participants with events | 5.3 [1.3 to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm A (Nivolumab Alone) vs Arm B (Nivolumab + Nab-Paclitaxel); Test type: Superiority; p = 0.5186, Log Rank

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Arm A (Nivolumab Alone) | Arm B (Nivolumab + Nab-Paclitaxel)
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Nivolumab Alone) (N=3) | Arm B (Nivolumab + Nab-Paclitaxel) (N=4)
Death NOS (General disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Nivolumab Alone) (N=3) | Arm B (Nivolumab + Nab-Paclitaxel) (N=4)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (5) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 2 (5)
Weight gain (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT02967133/Prot_SAP_000.pdf